CLINICAL TRIAL: NCT01218672
Title: A Prospective Multicenter Randomized Study Comparing Photoselective Vaporization of the Prostate With the GreenLight XPS™ Laser System and Transurethral Resection of the Prostate for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Photoselective Vaporization of the Prostate With the GreenLight XPS™ Laser System vs TURP for the Treatment of BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE1006
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GreenLight XPS (Experimental): Photoselective vaporization of the prostate using GreenLight XPS laser system.
  Interventions: Device: Photoselective Vaporization of the Prostate
- Transurethral Resection of the Prostate (Active Comparator): Monopolar and bipolar Transuretheral resection of the prostate (TURP)
  Interventions: Device: Transurethral Resection of the Prostate

INTERVENTIONS:
Device: Photoselective Vaporization of the Prostate — GreenLight XPS laser console GreenLight XPS consists of a 532 nm laser console capable of achieving power outputs between 20W and 180W. Laser technology is used to vaporize tissue for debulking prostatic hyperplasia and improvement of lower urinary tract symptoms. The 532 nm wavelength is in the visible spectrum as green light and is strongly absorbed by oxyhemoglobin.
  GreenLight XPS will be used in conjunction with the MoXy™ fiber. The fiber features a side firing mechanism delivering up to180W of 532 nm light to vaporize and coagulate the prostate tissue. The fiber is guided to the treatment site by the continuous flow cystoscope, consisting of an inner and outer sheath set, 30ْ forward oblique telescope and visual obturator.
  Arms: GreenLight XPS
Device: Transurethral Resection of the Prostate — Monopolar and bipolar loop TURP Systems The TURP procedure requires the use of a resectoscope, camera system and irrigation fluid. The system consists of a generator unit and a wire loop with an electrical current running through the loop used to cut prostate tissue and cauterize. Prostate tissue is cut away in small pieces and removed at the end of the procedure using irrigation. There are many manufacturers of TURP systems. Any monopolar and bipolar loop system that carry the CE mark may be used for the study.
  Arms: Transurethral Resection of the Prostate

SUMMARY:
The study compares procedural and post procedural outcomes for photoselective vaporization of the prostate (PVP) and transurethral resection of the prostate (TURP) for the treatment of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction. The study requires use of the CE marked GreenLight XPS™ Laser System (GreenLight XPS) or a CE marked monopolar or bipolar loop TURP system for the treatment of benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
The study will compare procedural and post procedural outcomes for photoselective vaporization of the prostate (PVP) and transurethral resection of the prostate (TURP) for the treatment of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction. The study requires use of the CE marked GreenLight XPS™ Laser System (GreenLight XPS) or a CE marked monopolar or bipolar loop TURP system for the treatment of benign prostatic hyperplasia (BPH). The purpose of the study is to demonstrate that PVP is not inferior to TURP.

ELIGIBILITY:
Inclusion criteria:

* Subject has provided informed consent and agrees to attend all study visits
* Subject has diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction
* Subject is willing to be randomized
* Subject is able to complete self-administered questionnaires
* Clinical investigator has documented in the subject's medical record that in his/her judgment the subject is a surgical candidate for either the PVP or the TURP procedure and may be randomized into either arm
* Subject is 40 to 80 years of age
* Subject has an IPSS score greater than or equal to 12 measured at the baseline visit
* Subject has medical record documentation of a maximum urinary flow rate (Qmax) less than 15ml/s (If uroflow testing documentation is available within 90 days prior to the informed consent date, and the sample is greater than or equal to 150ml, and the Qmax is less than 15ml/s it may be used for the inclusion/exclusion criteria)
* Subject has medical record documentation of a prostate volume of less than or equal to 100g by transrectal ultrasound (TRUS) (If TRUS testing documentation is available from less than 180 days prior to the informed consent date and the prostate volume is less than or equal to 100g, it may be used for the inclusion/exclusion criteria)
* Subject is classified as American Society of Anesthesiologists (ASA) I, II or III
* Subject has a serum creatinine that is within the normal range for the laboratory at the study center (or documentation of clinical insignificance in the subject's medical record by the investigator if outside the normal range) and measured less than or equal to 30 days prior to the date of surgery.

Exclusion criteria:

* Subject has a life expectancy of less than 2 years
* Subject is currently enrolled in, or plans to enroll in, any concurrent drug or device study unless preapproved by the sponsor
* Subject has an active infection (eg, urinary tract infection or prostatitis)
* Subject has a diagnosis of, or has received treatment for, chronic prostatitis or chronic pelvic pain syndrome (eg, non-bacterial chronic prostatitis)
* Subject has been diagnosed with a urethral stricture or bladder neck contracture within the 180 days prior to the informed consent date
* Subject has been diagnosed with 2 or more urethral strictures and/or bladder neck contractures within the 5 years prior to the informed consent date
* Subject has a diagnosis of lichen sclerosus
* Subject has a neurogenic bladder or other neurological disorder that would impact bladder function (eg, multiple sclerosis, Parkinson's disease, spinal cord injuries)
* Subject has a diagnosis of polyneuropathy (eg, diabetic)
* Subject has history of lower urinary tract surgery (eg, TURP, laser, urinary diversion, artificial urinary sphincter, penile prosthesis)
* Subject has diagnosis of stress urinary incontinence that requires treatment or daily pad/device use
* Subject has a history of intermittent self catheterization
* Subject has been catheterized or has a PVR >400mls in the 14 days prior to the surgical procedure
* Subject has current diagnosis of bladder stones
* Subject has diagnosis of prostate cancer
* Subject has a history of CIS, TaGII, TaGIII or any T1 stage bladder cancer
* Subject has damage to external urinary sphincter
* Subject has a medical contraindication for undergoing either TURP or PVP surgery (eg, infection, coagulopathy or significant cardiac or other medical risk factors for surgery)
* Subject has a disorder of the coagulation cascade (eg, hemophilia) or disorders that affect platelet count or function (eg, Von Willebrand's disease) that would put the subject at risk for intraoperative or postoperative bleeding
* Subject is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (3-5 days) except for low dose aspirin (eg, less than or equal to 100mg)
* Subject has had an acute myocardial infarction, open heart surgery or cardiac arrest less than 180 days prior to the date of informed consent
* Subject is immunocompromised (eg, organ transplant, leukemia)

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2011-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bachman, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland; Andrew Thomas, MBBCh, FRCS, Principal Investigator — Princess of Wales Hospital, Bridgend Mid Glamorgan
Locations (29):
- Krankenhaus der Barmherzigen Schwestern Linz, Linz, Austria
- AZ Maria Middelares Gent, Ghent, Belgium
- France (2):
  - Nouvel Hopital Civil de Strasbourg, Strasbourg
  - CHU Bretonneau, Tours
- Germany (9):
  - Campus Bejamin Franklin Hindenburgdamm, Berlin
  - UroForshungs GmbH, im St. hedwig Krankenhaus, Berlin
  - Krankenhaus Nordwest, Frankfurt
  - University Hospital of Heidelberg, Heidelberg
  - Hospital University of Jena, Jena
  - Universitatsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitatsklinikum Leipzig, Leipzig
  - Universitatsklinikum Magdeburg, Magdeburg
  - Diakoniekrankenhaus Rotenburg (W.) gGmbH, Rotenburg (Wümme)
- Unita di chirurgia Urologica mininvasiva,Azienda Ospedatiera Sant'Andrea Hospital, Rome, Italy
- Netherlands (2):
  - ZGT Almelo, Almelo
  - RadBound University Njmegen Medical Centre, Nijmegen
- Spain (2):
  - Hospital Iniversitario Fundacion Alcorcon, Madrid
  - Hospital de Manacor, Manacor
- University of Basel, Basel, Switzerland
- United Kingdom (10):
  - Frimley Park Hospital, Frimley, Camberley Surrey
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, Hampshire
  - Princess of Wales Hospital, Mid Glamorgan, Wales UK
  - Mid Yorkshire NHS Trust Dewsbury & District Hospital, Dewsbury
  - Western General Hospital, Edinburgh
  - Kent and Canterbury Hospital, Kent
  - Kings's College Hospital, London
  - Whipps Cross University Hospital, London
  - Freeman Hospital, Newcastle

REFERENCES:
- [Derived] Thomas JA, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Bachmann A. A Multicenter Randomized Noninferiority Trial Comparing GreenLight-XPS Laser Vaporization of the Prostate and Transurethral Resection of the Prostate for the Treatment of Benign Prostatic Obstruction: Two-yr Outcomes of the GOLIATH Study. Eur Urol. 2016 Jan;69(1):94-102. doi: 10.1016/j.eururo.2015.07.054. Epub 2015 Aug 15. PMID 26283011
- [Derived] Bachmann A, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Thomas JA. 180-W XPS GreenLight laser vaporisation versus transurethral resection of the prostate for the treatment of benign prostatic obstruction: 6-month safety and efficacy results of a European Multicentre Randomised Trial--the GOLIATH study. Eur Urol. 2014 May;65(5):931-42. doi: 10.1016/j.eururo.2013.10.040. Epub 2013 Nov 11. PMID 24331152

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten subjects were determined to be ineligible for the study procedure and were withdrawn before randomization (i.e., study procedure not performed).
Groups:
- TURP: Monopolar and bipolar loop TURP Systems
Period: Overall Study
Arm/Group | GreenLight XPS | TURP
Started | 139 | 142
Treated | 136 | 133
Completed | 128 | 121
Not Completed | 11 | 21

BASELINE CHARACTERISTICS:
Groups:
- GreenLight XPS: Photoselective vaporization of the prostate using GreenLight XPS laser system.
  GreenLight XPS vs. TURP: GreenLight XPS laser console GreenLight XPS consists of a 532 nm laser console capable of achieving power outputs between 20W and 180W. Laser technology is used to vaporize tissue for debulking prostatic hyperplasia and improvement of lower urinary tract symptoms. The 532 nm wavelength is in the visible spectrum as green light and is strongly absorbed by oxyhemoglobin.
- TURP: Monopolar and bipolar Transuretheral resection of the prostate (TURP)
  The TURP procedure requires the use of a resectoscope, camera system and irrigation fluid. The system consists of a generator unit and a wire loop with an electrical current running through the loop used to cut prostate tissue and cauterize. Prostate tissue is cut away in small pieces and removed at the end of the procedure using irrigation. There are many manufacturers of TURP systems. Any monopolar and bipolar loop system that carry the CE mark may be used for the study.
- Total: Total of all reporting groups
Arm/Group | GreenLight XPS | TURP | Total
Number analyzed (Participants) | 136 | 133 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (6.8) | 66.7 (6.6) | 67.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 136 | 133 | 269
Region of Enrollment [Number; unit: participants who were treated]
  France | 8 | 7 | 15
  Spain | 8 | 8 | 16
  Belgium | 5 | 5 | 10
  Austria | 4 | 4 | 8
  Germany | 28 | 35 | 63
  Netherlands | 13 | 12 | 25
  Italy | 12 | 10 | 22
  Switzerland | 10 | 12 | 22
  United Kingdom | 48 | 40 | 88

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: The IPSS is a patient-administered 7-question instrument used to classify severity of benign prostatic hyperplasia symptoms (BPH). Total scores can range from 0 to 35 (asymptomatic to very symptomatic).
Time Frame: 6 months
Population: The analysis includes all subjects who received a study treatment and for whom the outcome measure is available. Subjects were analyzed according to treatment received (as-treated analysis).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 134 | 131
units on a scale | 6.8 (5.2) | 5.6 (4.9)

2. Secondary Outcome: Maximum Urinary Flow Rate (Qmax)
Description: Qmax measured from a void of at least 150 ml in volume.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/s
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 116 | 117
ml/s | 23.3 (10.1) | 24.3 (11.4)

3. Secondary Outcome: Freedom From Complications
Description: A complication is defined as a device or procedure-related adverse event meeting at least 1 of the following criteria: Perforation of tissue or a physiologic structure; Required a prolonged or secondary hospitalization; Required surgical or invasive intervention (e.g., breaking of the skin) and excluding urinary catheterization for transient retention lasting less than 7 days and/or IV medications related to anesthesia.
Time Frame: 180 days
Measure: Number; unit: percentage of patients complication free
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 134 | 132
percentage of patients complication free | 87.3 | 83.3

4. Secondary Outcome: Prostate Volume
Description: Prostate volume measured via transrectal ultrasound
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 132 | 127
ml | 23.0 (11.7) | 20.5 (11.7)

5. Secondary Outcome: Post Treatment Outcomes of PVP and TURP
Description: Short Form Health Survey (SF-36 Acute) collected at 3-week visit. The SF-36 is a multi-purpose, short-form, health survey of functional health and well-being scores in a three-section format: Utility Index (score = 0-1 with higher score being better); Physical Component Summary (PCS) comprising of physical functioning, role-physical, bodily pain, and overall general health; Mental Component Summary (MCS) comprising of vitality, social functioning, role-emotional, and mental health. Each component in the PCS and MCS sections have a score of 1-100 with the higher score being better. The acute version uses a 1-week recall period.
Time Frame: 3 weeks post treatment
Population: A total of 136 subjects underwent GL-XPS and 133 subjects underwent TURP procedures. The SF36 questionnaire is comprised of three sections; available data is:
  SF36 (PCS): 133 GL-XPS, 129 TURP; SF36 (MHS): 134 GL-XPS, 130 TURP; SF36 Utility Index: 125 GL-XPS, 121 TURP.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 136 | 133
score
  SF36 - PCS: number analyzed (Participants) | 133 | 129
  SF36 - PCS | 50.3 (8.1) | 50.5 (7.3)
  SF36 - MHS: number analyzed (Participants) | 134 | 130
  SF36 - MHS | 50.0 (9.7) | 50.0 (10.9)
  SF36 Utility Index: number analyzed (Participants) | 125 | 121
  SF36 Utility Index | 0.7 (0.1) | 0.7 (0.1)

6. Secondary Outcome: Immediate Post Treatment Outcomes of PVP and TURP
Description: Length of stay calculated as the difference from entering the recovery room date/time to discharge date/time
Time Frame: 3 weeks
Population: A total of 136 subjects underwent GL-XPS and 133 subjects underwent TURP procedures. Length of Stay data available for 134 GL-XPS and 132 TURP subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 134 | 132
hours | 65.5 (63.3) | 97.8 (63.4)

7. Secondary Outcome: Health Status of PVP and TURP
Description: The IPSS, OABq, SF-36 Health Summary and EQ-5D instruments will be scored. IPSS classifies voiding symptoms with scores from 0-35 (asymptomatic to very symptomatic). The OABq captures overactive bladder symptom bother with scores from 0-100 (lower score is better). The SF-36 is a health survey with scores from 1-100 (higher score is better). EQ-5D assesses health status across a range of conditions and treatments with a score of 0-1 (higher score is better).
Time Frame: Baseline and 24-months
Population: Table reflects available data at specified time-points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 136 | 133
units on a scale
  Baseline IPSS: number analyzed (Participants) | 136 | 132
  Baseline IPSS | 21.2 (5.9) | 21.7 (6.4)
  Baseline OABq: number analyzed (Participants) | 134 | 132
  Baseline OABq | 44.2 (20.5) | 42.9 (20.8)
  Baseline SF-36 Health Summary: number analyzed (Participants) | 133 | 133
  Baseline SF-36 Health Summary | 52.2 (7.8) | 51.9 (7.1)
  Baseline EQ5D: number analyzed (Participants) | 133 | 132
  Baseline EQ5D | 0.843 (0.193) | 0.823 (0.219)
  24-Month IPSS: number analyzed (Participants) | 127 | 121
  24-Month IPSS | 6.9 (6.0) | 5.9 (6.1)
  24-Month OABq: number analyzed (Participants) | 126 | 120
  24-Month OABq | 15.3 (16.7) | 11.9 (13.7)
  24-Month SF-36 Health Summary: number analyzed (Participants) | 127 | 120
  24-Month SF-36 Health Summary | 52.5 (8.1) | 53.2 (8.5)
  24-Month EQ5D: number analyzed (Participants) | 127 | 119
  24-Month EQ5D | 0.875 (0.194) | 0.857 (0.210)

8. Secondary Outcome: Tolerability of PVP and TURP Assessed Using International Index of Erectile Function (IIEF-5) and International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF)
Description: The International Index of Erectile Function (IIEF-5) and International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) instruments will be collected at baseline and the follow-up visits.
  The IIEF-5 is a self-administered 5 question instrument that assesses the relevant domains of male sexual function such as erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction with a total possible score of 5-25 (higher score is better).
  The ICIQ-SFis a self-administered 4-question tool designed for the assessment and quantification of incontinence and its impact on quality of life during the previous 4 weeks with a total score of 0-21 (higher score is worse).
Time Frame: Baseline, 12-months, and 24-months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GreenLight XPS: Photoselective vaporization of the prostate using GreenLight XPS laser system.
  Photoselective Vaporization of the Prostate: GreenLight XPS laser console GreenLight XPS consists of a 532 nm laser console capable of achieving power outputs between 20W and 180W. Laser technology is used to vaporize tissue for debulking prostatic hyperplasia and improvement of lower urinary tract symptoms. The 532 nm wavelength is in the visible spectrum as green light and is strongly absorbed by oxyhemoglobin.
  GreenLight XPS will be used in conjunction with the MoXy™ fiber. The fiber features a side firing mechanism delivering up to180W of 532 nm light to vaporize and coagulate the prostate tissue. The fiber is guided to the treatment site by the continuous flow cystoscope, consisting of an inner and outer sheath set, 30ْ forward oblique telescope and visual obturator.
Arm/Group | GreenLight XPS | Transurethral Resection of the Prostate
Number analyzed (Participants) | 136 | 133
units on a scale
  Baseline IIEF-5 | 13.2 (7.6) | 13.7 (7.5)
  Baseline ICIQ-UI SF | 3.9 (4.7) | 4.4 (4.6)
  24-Months IIEF-5 | 12.9 (7.5) | 13.9 (8.2)
  24-Months ICIQ-UI SF | 2.8 (4.1) | 2.0 (3.3)

9. Secondary Outcome: Subject Satisfaction of PVP and TURP
Description: Subject responses to satisfaction with treatment as collected on follow-up visits.
  Data presented below indicates responses from subjects that would go through study treatment again at each of the defined follow-up visits.
Time Frame: 3-weeks, 3-months, 6-months, 12-months, and 24-months
Population: Descriptive statistics including frequency and percentages will be calculated. Results presented below are number of respondents who said Yes.
Measure: Count of Participants; unit: Participants
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 125 | 120
Participants | 116 | 107

10. Secondary Outcome: Rate of Retreatment of PVP and TURP
Description: Subject experiencing a retreatment (removal of tissue via TUPR, PVP, or other intervention) for obstruction after the initial procedure was required
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | GreenLight XPS | TURP
Number analyzed (Participants) | 136 | 133
Participants
  Months 0-6 | 4 | 7
  Months 7-12 | 6 | 2
  Months 13-24 | 4 | 1

ADVERSE EVENTS:
Time Frame: From the date of the informed consent until the subject exits the study. (Mean follow-up was 23.3 months)
Description: Adverse events determined as "Other" were not further defined during analysis.
Groups:
- TURP: Monopolar and bipolar Transuretheral resection of the prostate (TURP)
Arm/Group | GreenLight XPS | TURP
Serious Adverse Events (participants affected / at risk) | 24/136 | 25/133
Other Adverse Events (participants affected / at risk) | 68/136 | 57/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GreenLight XPS (N=136) | TURP (N=133)
Bleeding (Renal and urinary disorders) | 3 (3) | 8 (9)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3) | 2 (2)
Irritative symptoms/pain/discomfort (Renal and urinary disorders) | 1 (1) | 0 (0)
Stricture (Renal and urinary disorders) | 8 (8) | 7 (7) — meatal, urethral, bladder neck
Urinary Incontinence (Renal and urinary disorders) | 6 (7) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 5 (5) | 6 (6)
Other (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GreenLight XPS (N=136) | TURP (N=133)
Bleeding (Vascular disorders) | 13 (13) | 13 (13)
Urinary Tract Infection (Renal and urinary disorders) | 25 (26) | 12 (14)
Irritative Symptoms/Pain/Discomfort (Renal and urinary disorders) | 30 (33) | 30 (30)
Stricture (meatal, urethral, bladder neck) (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary Incontinence (Renal and urinary disorders) | 10 (10) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 13 (13) | 9 (9)
Other (Renal and urinary disorders) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No